CLINICAL TRIAL: NCT01254682
Title: Intra-articular Hyaluronan Substitution in Arthroscopy of the Wrist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TRB Chemedica AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSTWA-07-01
Record Dates: First submitted 2010-11-22; First posted 2010-12-06 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Arthroscopic Surgery
Keywords: wrist; joint; arthroscopy; hyaluronan; hyaluronic acid; Necessity of Arthroscopic surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyaluronic acid sodium salt (1%, 20mg/2ml) (Active Comparator)
  Interventions: Device: Ostenil
- Standard arthroscopic procedure (Other)
  Interventions: Procedure: Standard arthroscopic procedure

INTERVENTIONS:
Device: Ostenil — Standard arthroscopy (including intra-articular injection of 5 ml scandicain (0,5%), or 5 ml bupivacain plus 5 ml suprarenin in case of post-arthroscopic treatment). Add-on treatment with Ostenil after standard arthroscopic procedure. Application twice: first injection directly after arthroscopic procedure and second injection 3 weeks post arthroscopic.
  Arms: Hyaluronic acid sodium salt (1%, 20mg/2ml)
Procedure: Standard arthroscopic procedure — Standard arthroscopy (including intra-articular injection of 5 ml scandicain (0,5%), or 5 ml bupivacain plus 5 ml suprarenin in case of post-arthroscopic treatment) without add-on treatment.
  Arms: Standard arthroscopic procedure

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of Ostenil application (1% hyaluronan) after arthroscopy of the wrist.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 80 years of age
* Minimum pain score of 2 according to modified Mayo Wrist Score
* Patients in good general health/nutritional condition
* Signed written informed consent

Exclusion Criteria:

* Alcohol / drug abuse, drug addiction or neurotic personality disorder; patients with mental illness or suicidal tendency
* Severe intercurrent illness (like uncontrolled diabetes mellitus or thyroid disease, carcinoma,...)
* Fertile women without medically secured contraception(hysterectomy, sterilization, contraceptives,...)
* Subjects having a high probability of non compliance to the study procedures according to investigator's judgement (like illiteracy, insufficient German linguistic knowledge)
* Contraindication for the use of one of the investigational products or for the scheduled anesthesia
* Concomitant or previous participation in a clinical trial within the last 3 months
* Intraarticular treatment with a sodium hyaluronate-based product within the last 6 months
* Intraarticular treatment by the use of corticoid containing substance within the last 3 months
* Concomitant illness or injury influencing study evaluation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Inter-group comparison of Mayo total wrist score in subjects with or without post-arthroscopic hyaluronan treatment 3 months after arthroscopic surgery. | Baseline and 3 months
  Mayo wrist score evaluation consisting of 4 sections:
  * Maximal grip strength on injured side (compared to maximal strength of contralateral side, measured by 4-point scale, ranking from '0' for minimal to '30' for maximal strength)
  * Range of motion (measured by 4-point scale, ranking from '0' for minimal to '20' for maximal mobility)
  * Pain (measured by 4-point scale, ranking from '0' for maximal to '20' for minimal pain)
  * Function in daily activities (measured by 4-point scale, ranking from '0' for minimal to '30' for maximal function)

SECONDARY OUTCOMES:
Inter-group comparison of Mayo total wrist score in subjects with or without post-arthroscopic hyaluronan treatment. | Measured during the 6-month duration of participation
Disabilities of the arm, shoulder, and hand (DASH) outcome measure | Measured during the 6-month duration of participation
Grip strength | Measured during the 6-month duration of participation
Visual analogue scale of pain (VAS; 100 mm) | Measured during the 6-month duration of participation
Clinical Global Impression (CGI) | Measured during the 6-month duration of participation
Inter-group comparison of Mayo wrist subscores in subjects with or without post-arthroscopic hyaluronan treatment. | Measured during the 6-month duration of participation
  * Maximal grip strength on injured side (compared to contralateral side)
  * Range of motion
  * Pain
  * Function in daily activities
Number of subjects with Adverse Events as a measure of safety and tolerability | Measured during the 6-month duration of participation

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Schütz, Dr. med., Principal Investigator — Orthopädische Gemeinschaftspraxis, Straubing (Germany)
Locations (1):
- Orthopädische Gemeinschaftspraxis, Straubing, Bavaria, Germany